CLINICAL TRIAL: NCT00125567
Title: Multicentre, Randomised, Double-Blind Study to Compare Stalevo to Levodopa/Carbidopa in Patients With Parkinson's Disease Experiencing Symptoms of Early Wearing-Off
Brief Title: Stalevo in Early Wearing-Off Patients
Acronym: SEWOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Andrew Wighton, Orion Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2939111; EudraCT number: 2004-005234-39
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo; Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stalevo (levodopa/carbidopa/entacapone)
  Interventions: Drug: Stalevo (levodopa/carbidopa/entacapone)
- 2 (Active Comparator): Levodopa/carbidopa
  Interventions: Drug: Levodopa/carbidopa

INTERVENTIONS:
Drug: Stalevo (levodopa/carbidopa/entacapone) — Oral, 50-150 mg levodopa four times daily, for up to 2 years
  Arms: 1
Drug: Levodopa/carbidopa — Oral capsules, 50-150 mg levodopa four times daily, for up to 2 years
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate in patients with Parkinson's disease that, when compared to levodopa/carbidopa, Stalevo will delay the time from initiation of study drug to the time an increase in antiparkinsonian medication is required due to inadequately controlled parkinsonian symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Treatment with 3 equal daily doses of levodopa/carbidopa up to 450 mg/day
* Unchanged antiparkinsonian medication for 6 weeks prior to baseline

Exclusion Criteria:

* Secondary or atypical parkinsonism
* Patients with daily unpredictable OFF periods or painful dyskinesia

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The time until a patient requires changes in antiparkinsonian therapy due to inadequately controlled parkinsonian symptoms | Up to 2 years of treatment

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Up to 2 years of treatment
Clinical Global Impression of Change (investigator) | Up to 2 years of treatment
Parkinson's Disease Questionnaire (PDQ-39) | Up to 2 years of treatment
Work Impairment Questionnaire | Up to 2 years of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wighton, BSc (Hons), Study Director — Orion Corporation, Orion Pharma; Bhadravati SD Sastry, FRCP, Principal Investigator — University Hospital of Wales and Rookwood Hospital
Locations (19):
- Denmark (3):
  - Aalborg Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Århus Kommunehospital, Nørrebrogade 44
- Finland (2):
  - South Karelia Central Hospital, Lappeenranta
  - Tampere University Hospital, Tampere
- Germany (5):
  - Parkinson Klinik Bad Nauheim, Bad Nauheim
  - Neurologische Klinik Bad Neustadt, Bad Neustadt an der Saale
  - Neurologische Klinik der Universitat Dusseldorf, Düsseldorf
  - Allgemeines Krankenhaus Harburg, Hamburg
  - Praxis Drs Lang, Krauss, Schreiber, Ulm
- Mater Private Hospital, Dublin, Ireland
- Sweden (2):
  - Universitetssjukhuset MAS, Malmo
  - Läkarhuset Vällingby, Vällingby
- United Kingdom (6):
  - Movement Disorder Services, Chertsey, Surrey
  - University Hospital of Wales, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Wales
  - Frenchay Hospital, Bristol
  - Leigh Infirmary, Leigh
  - Southampton General Hospital, Southampton